CLINICAL TRIAL: NCT04936919
Title: Pilot Evaluation of Smart vs HERO Broadband Light Treatment for Pigmented Skin Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBLCIP002
Record Dates: First submitted 2021-06-21; First posted 2021-06-23 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Pigmented Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects in the treatment arm will receive broadband light treatment
  Interventions: Device: BroadBand Light

INTERVENTIONS:
Device: BroadBand Light — Treatment arm will receive Broadband light treatment

SUMMARY:
The purpose of the study is to investigate the effects of Intense Pulsed Broad Band Light for treatment of pigmented lesions

DETAILED DESCRIPTION:
This study is conducted to investigate the effects of intense pulsed broadband light device for treatment of pigmented lesions

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, 18 years or older
* Fitzpatrick skin type I-III
* Has visible signs of moderate to severe skin pigmentation
* Willing to not use any other procedure(s) in the treatment area during the study, such as laser- or light-based treatment, non-light-based device treatment such as radiofrequency or ultrasound, injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler, chemical peel, or surgical procedure
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant or to father a child for the duration of the study
* Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes
* Subject must agree to not make any changes in their skin regimen for the duration of the study, including the follow-up period
* Subject must be able to read, understand and sign Informed Consent Form
* Must be willing to adhere to the treatment and follow-up schedule and post-treatment care instructions

Exclusion Criteria:

* Fitzpatrick skin type IV-VI
* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* Any type of prior cosmetic treatment to the target area within 3 months of study participation, such as laser or light-based procedures or surgery.
* Prior injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler in the target area within 1 week of study participation.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of retinoid, such as isotretinoin, or corticosteroid, as applicable, within 6 months of study participation.
* Topical use of retinoid, such as isotretinoin, corticosteroid or hydroquinone on the target area within 1 month of participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated, or unable/unlikely to refrain from tanning during the study (for example, subject's occupation requires regular sun exposure).
* Current smoker or history of smoking within 6 months of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Degree of improvement in photographs | 4 weeks
  photographs

CONTACTS AND LOCATIONS:
Overall Officials: Swengel, MD, Principal Investigator — RefinedMD
Locations (1):
- RefinedMD, Los Gatos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided